CLINICAL TRIAL: NCT03408379
Title: Impact of Platelet Activation in Intracranial Aneurysm Rupture Risk - PLAQRAN
Acronym: PLAQRAN
Status: Active, not recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: MMI_2017_27
Record Dates: First submitted 2018-01-17; First posted 2018-01-24 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Intracranial Aneurysms; Ruptured Aneurysm
Keywords: intracranial aneurysms; ruptured aneurysm; platelet activity
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm, Ruptured | interventions — Vasodilation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Collection of blood sample in aneurysm — In case of an endovascular treatment :
  * A blood sample (venous or arterial) of 10 ml will be taken at the beginning of the procedure, an intra aneurysmal blood sample (1mL) will be taken during the procedure and a blood sample (arterial) of 1 mL will be taken at the end of the procedure.
  * Iterative blood samples (arterial) of 10 mL will be taken at each follow up visit.
  In case of a surgery treatment :
  * A blood sample (venous or arterial) of 10 ml will be taken at the beginning of the surgery.
  * A Tissue sample will be taken during the surgery
  * Iterative blood samples (arterial) of 10 mL will be taken at each follow up visit.

SUMMARY:
Sub arachnoid hemorrhage consecutive to intracranial aneurysm rupture is a devastating disease. Predictors of intracranial aneurysm rupture are limited and focus mainly on size and location. Platelet activation may have a deleterious role on aneurysm rupture. The assumption is that patients with ruptured intracranial aneurysm will present a higher rate of platelet activation compared to patients with non ruptured aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 and over
* Patient presenting a single or multiple aneurysm
* Patient presenting an intracranial aneurysm for which an intervention is planned (endovascular treatment or surgery) : elective intervention for an unruptured aneurysm or emergency surgery for a broken aneurysm

Exclusion Criteria:

* Pregnant or breast feeding woman
* Patient benefiting from legal protection measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting a single or multiple intracranial aneurysm for which an intervention is planned (endovascular treatment or surgery)
Sampling Method: Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2032-06-23 (Estimated); Study Completion 2033-06-23 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with platelet activation | in the 7 days before embolisation
  comparison of this proportion between patients with ruptured versus non ruptured intracranial aneurysm

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique A. de Rothschild, Paris, France, France